CLINICAL TRIAL: NCT01997346
Title: Multi-level Determinants of Late ART Initiation in Sub-Saharan Africa (LSTART Study): A Cross-sectional Qualitative Situation Analysis at 4 HIV Care and Treatment Clinics in Ethiopia
Brief Title: Multi-level Determinants of Starting ART Late: Aim 2
Acronym: LSTART
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Batya Elul, Assistant Professor of Clinical Epidemiology, Columbia University
Other Study IDs: AAAI1192; 1R01MH089831 (NIH)
Record Dates: First submitted 2013-11-08; First posted 2013-11-28 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Human Immunodeficiency Virus (HIV); Acquired Immune Deficiency Syndrome (AIDS)
Keywords: ART initiation; Ethiopia; Clinic observation; VCT observation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Key Informant Interviews: We will conduct interviews with 4 clinic personnel (16 across the 4 sites) to learn about practices and provider perspectives in the HIV clinic or ancillary clinics such as VCT. The 4 clinic personnel in each site will include: the physician-in-charge, a nurse, one peer educator, and a nurse or community counselor from the VCT clinic. A semi-structured interview guide will be used to query respondents about: procedures for enrolling new clients, conducting active testing, identifying and initiating patients on ART, CD4 monitoring, tracking clients who have missed appointments, support programs, and peer education. We will also aim to understand how each respondent views her/his role, how s/he counsels patients on pre-ART care, and the challenges faced from each one's perspective.

SUMMARY:
The availability of HIV care and treatment programs is increasing in sub-Saharan Africa. However more than half the patients who need HIV medicines are still not receiving this antiretroviral therapy (ART), and this can lead to early death from AIDS. One of the problems in this region is that patients start ART late, after the HIV disease is very advanced. This results in high death rates soon after ART initiation. The way clinic-level factors, such as the way services and referrals are organized, how referrals are regarded, counseling messages and record-keeping, contribute to late ART initiation is unclear. As the second phase of a 3-phase NIH-sponsored project, this study will identify clinic-level enablers and barriers to timely enrollment into HIV care and ART initiation. A cross-sectional qualitative study will be conducted at 4 selected HIV care and treatment clinics and the health facilities in which they are located in Ethiopia. Data will be collected using 4 methods:

1. Data abstraction
2. Key informant interviews with clinic personnel
3. Observation of post-test counseling sessions in the VCT clinic
4. Observation of provider-patient interactions in the care and treatment clinic Identifying modiﬁable health facility-level predictors of late ART initiation will facilitate implementation of interventions, programs and policies that will increase the number of patients who enroll in HIV care and initiate ART early. Additionally, results will inform the design of the third phase of the NIH-project referenced above.

DETAILED DESCRIPTION:
Background: Although HIV care and treatment programs are scaling up in sub-Saharan Africa, more than 50% of patients who need ART are not receiving it and signiﬁcant mortality from AIDS persists. One major challenge in this region is high rates of late ART initiation (i.e., in the advanced stages of HIV disease) which results in high rates of mortality soon after ART initiation. The clinic-level factors that contribute to late ART initiation are unclear.

Objective: As the second of a 3-phase NIH-sponsored project, this study aims to identify clinic-level enablers and barriers to timely ART initiation.

Methods: A cross-sectional qualitative study will be conducted at 4 purposively selected HIV care and treatment clinics in Ethiopia. Data will be collected using 4 methods:

1. Data abstraction
2. Key informant interviews with clinic personnel
3. Observation of post-test counseling sessions at the voluntary counseling and testing (VCT) clinic
4. Observation of provider-patient interactions in the care and treatment clinic Descriptive statistics will be produced from the data abstraction. Content analysis of key informant interviews will be conducted. Descriptive summaries will be produced from observations. All analyses will focus on identifying within- and across-clinic themes, and include triangulation across data collection methods to identify clinic-level enablers and barriers to timely ART initiation.

Expected use of results: Identifying modiﬁable clinic-level enablers and barriers to timely ART initiation will facilitate implementation of interventions, programs and policies to reduce late ART initiation. Additionally, results will inform the third phase of the NIH-project referenced above.

ELIGIBILITY:
The inclusion and exclusion criteria for the clinics and the various study participants are given below:

1. Data abstraction

   Inclusion criteria: N/A - all study sites included. Exclusion criteria: N/A - all study sites included. .
2. Key informant interviews

   Inclusion criteria:
   * ≥18 years of age;
   * paid or voluntary employee in the 4 study sites for ≥6 months;
   * and give verbal informed consent.

   Exclusion criteria:
   * <18 years of age;
   * employed at the 4 study sites <6 months;
   * and/or not willing to give verbal consent.
3. Observation of post-test counseling sessions in the VCT clinic

   Inclusion criteria:
   * Providers: ≥18 years of age; paid or voluntary employee in the 4 study sites for ≥6 months; responsible for HIV post-test counseling in VCT or PICT in the adult outpatient clinic; and give verbal informed consent
   * Patients: ≥18 years of age; unaware of HIV status, and give verbal informed consent.

   Exclusion criteria:
   * Providers: <18 years of age; employed <6 months; and/or not willing to give verbal consent.
   * Patients: <18 years of age; and/or not willing to give verbal consent.
4. Observation of provider-patient interactions in the care and treatment clinic

Inclusion criteria:

* Providers: ≥18 years of age; paid or voluntary employee in the care and treatment clinic of 4 study sites for ≥6 months; and give verbal consent.
* Patients: ≥18 years of age; not yet on ART (regardless of eligibility), receiving counseling or another service from one of the observed providers, and give verbal informed consent.

Exclusion criteria:

* Providers: <18 years of age; employed <6 months; and/or not willing to give verbal consent.
* Patients: <18 years of age; and/or not willing to give verbal consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will conduct key informant interviews with 4 clinic personnel (16 across the 4 sites) to learn about actual practices and provider perspectives in the HIV clinic or ancillary clinics such as VCT. The 4 clinic personnel in each site will include: the physician-in-charge of the HIV clinic, a nurse working in the HIV clinic, one peer educator from the HIV clinic, and a nurse or community counselor from the VCT clinic.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Percentage of provider-patient interactions that were observed to be rushed by visit type | 12 months
  Visit type includes post-test counseling, enrollment, 1st CD4, pre-ART monitoring, and ART preparatory.

CONTACTS AND LOCATIONS:
Overall Officials: Batya Elul, PhD, MSc, Principal Investigator — ICAP-NY, Columbia University
Locations (4):
- Ethiopia (4):
  - Fitche Hospital, Fichē
  - Goba Hospital, Goba
  - Nekemte Hospital, Nekemte
  - Shashemene Hospital, Shashemenē